CLINICAL TRIAL: NCT01627964
Title: Motion Analysis and Assessment of Cardiac Function for Cardiac Images
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yu-Chien Shiau, Physician, Far Eastern Memorial Hospital
Other Study IDs: FEMH-IRB-100070-E
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Heart; Functional Disturbance
Keywords: Heart Wall Motion Function

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- normal heart function: normal heart function
- abnormal heart function: abnormal heart function

SUMMARY:
The study develops software for motion analysis and assessment of cardiac function for cardiac images. Cardiac catheterization ventriculography of several randomly selected patients were taken from our hospital's PACS system. The investigators remove the patient information on the images, and use the image for motion analysis and assessment.

DETAILED DESCRIPTION:
The study develops software for motion analysis and assessment of cardiac function for cardiac images. Twenty patients who have both cardiac catheterization ventriculography and cardiac echo studies will be randomly selected. Cardiac catheterization ventriculography of the selected patients were taken from our hospital's PACS system. The investigators remove the patient information on the images, and use the image for motion analysis and assessment. The results will be compared and correlated with their cardiac echo, which could validate the clinical usefulness of the software.

ELIGIBILITY:
Inclusion Criteria:

* patients who already have cardiac catheterization ventriculography and cardiac echo studies.

Exclusion Criteria:

* patients who do not have either cardiac catheterization ventriculography or cardiac echo studies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: randomly selected patients
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chien Shiau, PhD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Bravo A, Medina R. An unsupervised clustering framework for automatic segmentation of left ventricle cavity in human heart angiograms. Comput Med Imaging Graph. 2008 Jul;32(5):396-408. doi: 10.1016/j.compmedimag.2008.03.003. PMID 18502609
- [Background] White RD, Setser RM. Integrated approach to evaluating coronary artery disease and ischemic heart disease. Am J Cardiol. 2002 Nov 21;90(10C):49L-55L. doi: 10.1016/s0002-9149(02)02964-8. PMID 12459428
- [Background] Oost E, Koning G, Sonka M, Oemrawsingh PV, Reiber JH, Lelieveldt BP. Automated contour detection in X-ray left ventricular angiograms using multiview active appearance models and dynamic programming. IEEE Trans Med Imaging. 2006 Sep;25(9):1158-71. doi: 10.1109/tmi.2006.877094. PMID 16967801
- [Background] Suzuki K, Horiba I, Sugie N, Nanki M. Extraction of left ventricular contours from left ventriculograms by means of a neural edge detector. IEEE Trans Med Imaging. 2004 Mar;23(3):330-9. doi: 10.1109/TMI.2004.824238. PMID 15027526